CLINICAL TRIAL: NCT07076498
Title: Phase 1 Trial of Engineered HSV-1 M032 in Children and Adults With Newly Diagnosed Diffuse Midline Glioma After Standard of Care Radiation
Brief Title: Engineered HSV-1 M032 for the Treatment of Children and Adults With Newly Diagnosed Diffuse Midline Glioma After Standard of Care Radiation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0876; CDMRP-PC250876 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2025-07-15; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Glioma
Keywords: Diffuse Midline Glioma; H3 K27-altered; H3 K27M-mutant; Pediatric Brain Tumor; DMG; Diffuse Intrinsic Pontine Glioma; Supratentorial DMG; DIPG; M032; Oncolytic Herpes Simplex Virus; Oncolytic Virus; oHSV; Immunotherapy; Oncolytic Immunotherapy; Viral Immunotherapy; Intratumoral Therapy; Phase 1 Trial; Pediatric Oncology; Neuro-Oncology; Clinical Trial in Children; Translational Research
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adult: For Adult Patients Phase 1 Treatment with Single Injection of M032 (Experimental): All patients in both disease cohorts (Cohort 1: Supratentorial DMG; Cohort 2: Pontine DMG) will be enrolled in this single-arm Phase 1 trial and will receive intratumoral administration of M032. Each patient will be treated with a single dose of M032 directly injected into the tumor. There is no placebo or comparator arm. The primary objectives are to evaluate the safety and tolerability of M032 and to determine the recommended Phase 2 dose (RP2D). The two disease cohorts will be assessed independently.
  Interventions: Biological: M032
- PED: For Pediatric Patients Phase 1 Treatment with Single Injection of M032 (Experimental): All patients in both disease cohorts (Cohort 1: Supratentorial DMG; Cohort 2: Pontine DMG) will be enrolled in this single-arm Phase 1 trial and will receive intratumoral administration of M032. Each patient will be treated with a single dose of M032 directly injected into the tumor. There is no placebo or comparator arm. The primary objectives are to evaluate the safety and tolerability of M032 and to determine the recommended Phase 2 dose (RP2D). The two disease cohorts will be assessed independently.
  Interventions: Biological: M032

INTERVENTIONS:
Biological: M032 — M032 is a genetically engineered type 1 herpes simplex virus (HSV-1) that has been demonstrated to be aneurovirulent secondary to deletions of both copies of the γ134.5 gene and modified to express human interleukin-12 (IL-12). Each patient will receive a single intratumoral injection of M032.

SUMMARY:
The goal of this clinical research study is to learn about the safety and effects of M032 given directly into the tumor in children and adults with DMG and who have received standard-of-care radiation therapy.

DETAILED DESCRIPTION:
Primary Objective:

I. To assess the safety and tolerability of IL-12-expressing HSV-1 NSC 733972 (M032) administered intratumorally via stereotactic intratumoral injection in children and adults with a diagnosis of diffuse midline glioma (DMG) after receiving standard of care radiation.To determine the maximum tolerated dose (MTD), which will serve as the recommended Phase 2 dose (RP2D). This will include two cohorts: supratentorial DMG H3K27-altered and pontine DMG.

Secondary Objective:

I. Obtain preliminary information concerning the potential efficacy of M032 by assessing longitudinal changes in radiographic response, progression free and overall survival, and performance scale.

II. To survey for virologic shedding in saliva, conjunctiva, and blood. III. To evaluate immunologic responses to M032 by assessing HSV antibody titers and changes from baseline in circulating peripheral blood immune cells, cytokines, and chemokines by longitudinal sampling.

Exploratory Objectives:

I. To evaluate pre- and post-treatment tissue for immune cell populations and checkpoint proteins in patients who are amendable to and meet criteria for resection/biopsy while on study.

II. To assess overall survival (OS) in subgroups of patients based on therapies received after M032 (surgery versus no surgery; reirradiation versus no reirradiation, immunotherapy versus [vs] no immunotherapy).

OUTLINE: This is a dose escalation study of M032.

Patients receive M032 intratumorally (IT) on day 0 over 5 minutes at the time of standard of care (SOC) craniotomy. Patients undergo magnetic resonance imaging (MRI), as well as saliva, conjunctival secretions, blood collection throughout the trial. Patients may undergo tissue biopsy on study.

After completion of study treatment, patients are followed up at 7, 14, and 28 days, then 3, 5, 7, 9, 12, 18, 24 and 36 months, and then annually up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 36 months
* Newly diagnosed pathologically proven diffuse midline glioma (DMG) (H3 K27M mutant) or radiographic and/or pathologically proven pontine DMG (tumors with an epicenter in the pontine and diffuse involvement in at least 50% of the axial diameter of the pons)
* Patient must have received standard of care radiation ≥ 4 but ≤ 8 weeks prior to study enrollment Note: The eligibility determination, enrollment, pre-surgical planning, and M032 administration must be completed within 8 weeks of radiation therapy completion.
* The tumor characteristics for enrollment are as follows:
* The lesion must be ≥ 1.0 cm and ≤ 4.0 cm in diameter and surgically accessible as determined by MRI
* For patients diagnosed with supratentorial DMG, tumors larger than 4.0 cm may be eligible if they can be surgically debulked to ≤ 4.0 cm
* Patients must have fully recovered from acute treatment-related toxicities prior to entering this study. The study entry timepoint is defined as the time of consent
* Previous treatment guidelines (if applicable):
* Monoclonal antibody (i.e., bevacizumab): patient must have received last dose ≥ 21 days prior
* Radiation: Patients must have received their last fraction of radiation ≥ 4 weeks and ≤ 8 weeks prior to study entry
* Temozolomide: Patients must have received their last dose of chemotherapy ≥ 4 weeks prior

Normal hematological, renal, and liver function as defined below:

* Hemoglobin > 9g/dL
* White blood cell ≥ 3,000/μL
* Absolute neutrophil count ≥ 1000/mm3
* Platelets ≥ 100,000/mm3
* PT or PTT ≤ 1.3 x control
* Creatinine within normal institutional limits OR creatinine clearance ≥ 60 mL/min/1.73 m2 (cystatin C preferred) for patients with creatinine levels above institutional normal
* Total Bilirubin ≤ 1.5 mg/dl
* Transaminases < 3 times above the upper limits of the institutional norm
* Patients < 16 years, Modified Lansky score ≥ 60; patients ≥ 16 years, Karnofsky score ≥ 60
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. (Refer to Pregnancy Assessment Policy MD Anderson Institutional Policy # CLN1114). This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:
* Postmenopausal (no menses in greater than or equal to 12 consecutive months).
* History of hysterectomy or bilateral salpingo-oophorectomy.
* Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
* History of bilateral tubal ligation or another surgical sterilization procedure.
* Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of study agent administration.
* Written informed consent in accordance with institutional and FDA guidelines must be obtained from the patient or legal guardian

Exclusion Criteria:

* Patients who previously received other investigational agents
* Patients with untreated symptomatic hydrocephalus
* Patients with a radiographic atypical pontine DMG or exophytic glioma, unless biopsy confirmed H3K27M alteration
* Patients with a primary spinal cord tumor
* Acute infection, granulocytopenia, or medical condition precluding surgery
* Pregnant or lactating females: Pregnant women are excluded from this study due to the unknown potential of M032 to cause teratogenic or abortifacient effects. Lactating females are excluded from this study due to the unknown potential risk of adverse effects on both the mother and nursing infants associated with treatment using M032
* Diagnosis of encephalitis or CNS infection < 12 weeks prior
* Receiving ongoing treatment for encephalitis, CNS infection, or multiple sclerosis
* Tumor involvement which would require ventricular inoculation or would require access through a ventricle to deliver treatment
* Patients may not be on immunosuppressive therapy (for at least 1 week), including corticosteroids at the time of enrollment. Physiological replacement of corticosteroids, intermittent use of bronchodilators, or topical steroids will not be excluded from the study.
* Known HIV seropositivity or known immune deficiency
* Patient with an active herpes infection with clinical symptomology
* Concurrent therapy with any drug active against HSV (acyclovir, valacyclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir) or any systemic immunosuppressive drug therapy (except physiological replacement of corticosteroids
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen for this trial.
* Concurrent anticancer or investigational drug
* Patients with medical contraindications for MRI or MRI contrast agents.
* Patients who have received a live vaccine within 30 days prior to planned M032 treatment.

Min Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kane Friedman Friedman, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org